CLINICAL TRIAL: NCT06687187
Title: Effect of Two Different Doses of Neostigmine on the Gastric Residual Volume and Aspiration in Critically Ill Patients Under Enteral Feeding; a Comparative Controlled Randomized Trial
Brief Title: Effect of Two Different Doses of Neostigmine on the Gastric Residual Volume and Aspiration in Critically Ill Patients
Acronym: Gastric
Status: Completed | Type: Observational
Sponsor: Zulekha Hospitals (Other)
Responsible Party: Sponsor
Other Study IDs: 382/46
Record Dates: First submitted 2024-11-10; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Gastric Reflux
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Neostigmine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group I: received neostigmine 1 mg
  Interventions: Drug: Neostigmine
- Group II: received neostigmine 2 mg
  Interventions: Drug: Neostigmine
- Group III: received normal saline

INTERVENTIONS:
Drug: Neostigmine — two groups (Group I, n= 41) and (Group II, n= 43) received varying doses of neostigmine (1 mg and 2 mg respectively
  Groups: Group I; Group II

SUMMARY:
A study comparing the effect of two doses of neostigmine on the gastric residual volume in critically ill patients on enteral feeding.

DETAILED DESCRIPTION:
Participants were categorized into three groups: Group I and Group II received neostigmine 1 mg and 2 mg, respectively, and a control group received 10 ml of normal saline. All participants received an intravenous administration of 10 mg of metoclopramide. GRV was measured every 3 hours before enteral feeding. aspiration through nasogastric (NG) or orogastric (OG) tubes was done before the next due bolus of feeding.

ELIGIBILITY:
Inclusion Criteria:

* patients with a GRV >120ml
* a normal heart rateExclusion Criteria
* absence of comorbidities such as diabetes and renal failure. exclusion Criteria:
* Patients exhibiting new-onset arrhythmias or heart block
* hypotension (systolic blood pressure less than 60 mmHg)
* experiencing active gastrointestinal bleeding or receiving prokinetic medications 8-12 hours before the intervention
* patients with a history of surgery in the gastrointestinal system in the past two weeks history of extrapyramidal manifestations
* patients with electrolyte imbalance
* pregnant patients,

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study included 124 patients aged between 20 and 60 years requiring enteral feeding via nasogastric (NG) or orogastric (OG) tubes
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
The risk of aspiration | december 2022 to may 2024
  The risk of aspiration in ICU patients on enteral feeding via vaso-gastric or oro-hastric tubes

CONTACTS AND LOCATIONS:
Overall Officials: abdalla e hassan, lecturer, Principal Investigator — lecturer
Locations (1):
- Al-Azhar faculty of medicine, Cairo, Egypt